CLINICAL TRIAL: NCT03224611
Title: Usefulness of Light Wand-guided Insertion of Flexible Reinforced Laryngeal Mask Airway: Comparison With Conventional Blind-insertion
Brief Title: Usefulness of Light Wand-guided Insertion of Flexible Reinforced Laryngeal Mask Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiyoung Yoo, clinical assistant professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AJIRB-MED-OBS-17-108
Record Dates: First submitted 2017-07-13; First posted 2017-07-21 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Laryngeal Mask Airway

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The flexible LMA is inserted using "index finger technique"
- Light wand group (Active Comparator): The flexible LMA is inserted using light wand as a stylet
  Interventions: Device: light wand

INTERVENTIONS:
Device: light wand — The light wand is used as a stylet of the flexible LMA. When the investigator inserts the flexible LMA in "light wand group", the correct position of the LMA is confirmed by the light.
  Arms: Light wand group

SUMMARY:
Flexible LMA (Laryngeal mask airway) is very useful for variable situation but it is hard to insert in correct position because of it's flexible structure. Especially in classical way of manual LMA insertion, when the index finger could not guide the flexible LMA to the optimal position, we could not guarantee the correct position of the LMA. Therefore several studies have been investigated to improve this.

The light wand is a kind of stylet which have a light on the tip. Recently some studies demonstrated the usefulness of the light wand which could be used for indicating correct position of the LMA. We hypothesised there will be two advantages if the light wand is used as a stylet of the flexible LMA. First the stylet could support the mildness of the flexible LMA, and second the lightness could confirm the correct position of the flexible LMA.

ELIGIBILITY:
Inclusion Criteria:

* The patient need general anesthesia using LMA and belonged to the ASA(American society of Anesthesiologist) class I or II

Exclusion Criteria:

* The patient who has URI(upper respiratory infection) symptom within 14 days or
* The patient's BMI(body mass index) exceeds 35 kg/m2
* The patient has severe GERD(gastroesophageal reflux disease) or hiatus hernia
* The patient who has any contraindication for LMA insertion

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Oropharyngeal leak pressure | 5 minutes after LMA is inserted
  The oropharyngeal leak pressure is measured by the pressure which the investigator could detect the audible sound by stethoscope on patient's cheek during the exhaust valve is closed and the fresh gas is allowed to flow into the lungs at 3 liters per minute.

SECONDARY OUTCOMES:
The grade of oropharyngeal view through the fiberoptic assessment | 5 minutes after LMA is inserted
  The position of the LMA was assessed by fiberoptic examination through an attachment between the LMA and the anesthetic circuit.

CONTACTS AND LOCATIONS:
Overall Officials: Ji Young Yoo, Principal Investigator — Clinical assistant professor
Locations (1):
- Ajou University Hospital, Suwon, Gyeonggido, South Korea

IPD SHARING:
Plan to Share IPD: No